CLINICAL TRIAL: NCT06616636
Title: A Phase Ib Study of Rezatapopt in Combination With Azacitidine in Patients With TP53Y220C Mutant Myeloid Malignancies (Acute Myeloid Leukemia or Myelodysplastic Syndrome)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (MSK) (Unknown); PMV Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0371; NCI-2024-08191 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rezatapopt + Azacitidine (Experimental): Participants will receive treatment on an inpatient or outpatient basis. Every cycle participants will take rezatapopt daily and receive azacitidine by IV for 7 days.
  Interventions: Drug: Azacitidine; Drug: Rezatapopt

INTERVENTIONS:
Drug: Azacitidine — Given by IV
Drug: Rezatapopt — Given orally with food

SUMMARY:
A non-randomized phase Ib study of PC14586 (PMV therapeutics) in patients diagnosed with TP53Y220C-mutant myeloid malignancies, including AML and MDS.

DETAILED DESCRIPTION:
Primary Objective:

To assess the safety and tolerability of rezatapopt in TP53Y220C -mutant myeloid malignancies (AML, MDS)

Secondary Objectives:

1. To determine the clinical efficacy of rezatapopt in R/R and newly diagnosed patients with TP53Y220C -mutant myeloid malignancies
2. To assess event free survival (EFS) and overall survival (OS) in patients receiving rezatapopt in combination with AZA +/- VEN
3. To assess duration of response in patients receiving rezatapopt in combination with AZA
4. Characterize the pharmacokinetics of rezatapopt in combination with AZA

Exploratory Objectives:

1. To assess changes in the variant allele frequencies of TP53Y220C mutations via next-generation sequencing.
2. To describe mutational profiles of patients on study at screening, response and at relapse and correlate to clinical parameters.
3. To assess changes in clonal architecture based on bone marrow aspirate samples using single cell sequencing.
4. To evaluate for p53 activation and changes in the immunologic profile of patients of TP53Y220C mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Patient is willing and able to adhere to the study visit schedule and other protocol requirements.
3. Patient has relapsed or primary refractory AML or MDS
4. Any other comorbidity that per the investigator renders a patient inappropriate for intensive chemotherapy.
5. Patients with MDS must be classified as MDS-IB1 or IB2 as per WHO 2022 criteria32
6. TP53Y220C mutation confirmed by CLIA-approved local testing with a variant allele frequency >2%.
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
8. Patient has adequate organ function defined as:

   * Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3 x ULN, unless considered due to leukemic organ involvement.
   * Serum total bilirubin ≤ 1.5 x ULN. Higher levels are acceptable if these can be attributed to ineffective erythropoiesis, leukemia organ involvement or Gilbert's syndrome.
   * Serum creatinine < 2 x ULN or creatinine clearance > 40 mL/min based on validated glomerular filtration rate (GFR) estimation (Cockcroft-Gault, CKD-epi, or MDRD equations).
9. Females of childbearing potential may participate provided they have a negative serum or urine pregnancy test at screening and a negative serum OR urine pregnancy test within 72 hours of starting on treatment. They also must agree to either abstain from sexual intercourse or use two forms of a highly effective method of contraception while on study and up to 3 months after the last dose of the study drug.
10. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) 14 days prior to study entry and for the duration of study participation. This includes all female patients between the onset of menses and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

    Postmenopausal (no menses in greater than or equal to 12 consecutive months). History of hysterectomy or bilateral salpingo-oophorectomy. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).

    History of bilateral tubal ligation or another surgical sterilization procedure.

    • Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

    Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of investigational agent administration.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patient has received prior chemotherapy, targeted therapy, immunotherapy, or treatment with an investigational anticancer agent within 14 days or 5 half-lives (if half-life is known), whichever is shorter, before receiving their first dose of study drug.
2. Patient has received radiotherapy within 14 days.
3. Patients with acute promyelocytic leukemia
4. Subject has immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
5. Patients with active, uncontrolled leukemia involvement of the CNS
6. Subject has known active viral infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
7. Subject is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
8. Subject has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
9. Patient has any unresolved toxicities from prior anti-cancer therapy greater than Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior chemotherapy induced neuropathy.
10. Patient has had major surgery within 2 weeks prior to the planned start of study treatment.
11. Female subject who is pregnant or lactating.
12. History of allergic reactions attributed to compounds of similar chemical or biologic composition to azacitidine, rezetapopt or other agents used in study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-08-27 (Estimated); Study Completion 2029-08-27 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Carter BZ, Mak PY, Ayoub E, Wu X, Ke B, Nishida Y, Futreal A, Ostermann LB, Bedoy AD, Boettcher S, DiNardo CD, Puzio-Kuter A, Poyurovsky MV, Levine A, Andreeff M. Restoring p53 wild-type conformation in TP53-Y220C-mutant acute myeloid leukemia. Blood. 2025 Nov 20;146(21):2574-2588. doi: 10.1182/blood.2025028935. PMID 40608889
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org